CLINICAL TRIAL: NCT07167537
Title: An Open-Label, Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Allogeneic CAR-T Cell Therapy (OL-CD19-GDT) in the Treatment of Relapsed/Refractory Autoimmune Diseases
Brief Title: A Study of OL-CD19-GDT in Relapsed/ Refractory Autoimmune Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Collaborators: Overland Therapeutics (Unknown)
Responsible Party: Principal Investigator, Jing Pan, Director of the department of Immunotherapy for Hematopoietic Malignancies, Beijing GoBroad Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OL-CD19-GDT-002
Record Dates: First submitted 2025-09-10; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Systemic Sclerosis (SSc); Primary Sjogren's Syndrome
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OL-CD19-GDT (Experimental)
  Interventions: Biological: OL-CD19-GDT

INTERVENTIONS:
Biological: OL-CD19-GDT — OL-CD19-GDT will be given through IV bolus with ascending dose levels to determine the RDE and RP2D as specified in the protocol

SUMMARY:
This study aims to characterize the safety, tolerability, pharmacokinetics, and preliminary efficacy of OL-CD19-GDT in relapsed/refractory autoimmune diseases.

DETAILED DESCRIPTION:
This is an open-label, single-arm, clinical study to evaluate the efficacy and safety of CAR-T therapy OL-CD19-GDT in the treatment of Relapsed/ Refractory Autoimmune Diseases such as SSc and pSS.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years old
* ECOG 0-2
* Adequate organ function
* Females of childbearing potential (FCBP) must have a negative pregnancy test at screening and must agree to use a highly effective contraceptive method starting from the time of lymphodepletion and for 2 years after dosing of the IMP
* SSc specific:

  a)Fulfilling the 2013 ACR/EULAR classification criteria of SSc; b) mRSS score >10; c) at least one vital organ involvement besides the skin; d)relapsed or refractory to at least one immunosuppressant or biologic.
* pSS specfic: a)Fulling the 2016 EULAR/ACR classification critieria for pSS; b) anti-Ro/anti-SSA antibody positive; c) ESSDAI score ≥5 ; d)relapsed or refractory to at least one immunosuppressant or biologic.

Exclusion Criteria:

* Active uncontrolled infection
* Serologic evidence of chronic hepatitis B virus (HBV) infection and unable or unwilling to receive standard prophylactic antiviral therapy or with detectable HBV viral load
* Serologic evidence of hepatitis C virus (HCV) infection without completion of curative treatment or with detectable HCV viral load
* HIV antibody positive
* Syphilis antibody positive
* Active tuberculosis, untreated or inadequately treated latent tuberculosis infection (LTBI)
* History of serious infection within 3 months prior to screening (defined as requiring hospitalization or intravenous antimicrobial therapy), or history of oral antimicrobial therapy within 1 month prior to screening (e.g., viral infections, opportunistic infections, including but not limited to severe cytomegalovirus or herpes virus infections)
* Congenital long QT syndrome or a corrected QTcF interval of ≥480 ms at screening (unless secondary to pacemaker or bundle branch block)
* Uncontrolled hypertension (blood pressure ≥160/100 mm Hg repeatedly), unstable angina, congestive heart failure (greater than New York Heart Association class II), electrocardiographic evidence of acute ischemia, coronary angioplasty or myocardial infarction within 6 months prior to screening, uncontrolled atrial or ventricular cardiac arrhythmia, poorly controlled diabetes or other endocrine diseases, severe chronic pulmonary disease, or other serious medical condition which is likely to significantly impair the patient's ability to tolerate the study treatment
* history of organ transplant
* Pregnancy or lactating women
* Use of any other experimental medication within 4 weeks or 5 half-lives prior to start of study drug
* Use of biologics within 10 weeks, stem cell transplant within 6 months prior to the start of study drug
* Prior CAR-T treatment
* Received live or attenuated vaccine within 4 weeks of Cycle 1 Day 1
* Presence of other autoimmune or auto-inflammatory diseases that may affect study assessments, such as rheumatoid arthritis, gout, or active fibromyalgia syndrome.
* Limited to patients diagnosed with SSc: at risk for scleroderma renal crisis; SSc-associated gastric antral vascular ectasia; Severe gastrointestinal involvement leading to malabsorption or intestinal failure
* Limited to patients diagnosed with pSS: primary biliary cholangitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | After OL-CD19-GDT administration up to 30 days (Day 1-Day 30)
  Adverse events will be assessed based on the CTCAE 5.0
Treatment emergent adverse event (TEAE) incidence and severity | From lymphodepletion through study completion, up to 2 years
  Adverse events will be assessed based on the CTCAE 5.0

SECONDARY OUTCOMES:
Overall Response Rate | Baseline through study completion, up to 2 years
  The efficacy outcome variable, Overall Response Rate (ORR), is defined as the ratio between the number of subjects experiencing a response at weeks 12, 24 and 52 and the total number of enrolled subjects. A response to treatment will be considered as:*SSc: Fulfillment of mCRISS criteria *pSS: Achieving ESSDAI response
Cmax of OL-CD19-GDT | Baseline through study completion, up to 2 years
  The maximum concentration of the CAR-T cells will be measured to assess OL-CD19-GDT in vivo expansion and persistence.
Tmax of OL-CD19-GDT | Baseline through study completion, up to 2 years
  The time of the maximum concentration will be measured to assess OL-CD19-GDT in vivo expansion and persistence.
AUC 0-28 days | Baseline through study completion, up to 2 years
  Area under the curve will be measured to assess OL-CD19-GDT in vivo expansion and persistence.
Serum cytokines | From lymphodepletion till day 90
  The levels of cytokines will be measured, such as IL-6.
Level of Immunogenicity | Baseline through study completion, up to 2 years
  To assess the presence of antibodies to OL-CD19-GDT (ADA)
Level of RCR | Baseline through study completion, up to 2 years
  To determine whether Replication Competent Retrovirus (RCR) is present in patients that receive OL-CD19-GDT

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing GoBroad Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No